CLINICAL TRIAL: NCT04706351
Title: The Arabic Version of Identification of Functional Ankle Instability Questionnaire(IdFAI-Ar)
Brief Title: Arabic Version of Identification of Functional Ankle Instability Questionnaire
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Aya Abdelhamied Mohamed Khalil, Lecturer of Kinesiology, Cairo University
Other Study IDs: P.T REC/012/001829
Record Dates: First submitted 2021-01-10; First posted 2021-01-12 (Actual); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Assessment
Keywords: Arabic; questionnaire; ankell instability

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: IdFAI questionnaire — The Identification of Functional Ankle Instability (IdFAI) is a newly published questionnaire that was specifically designed to detect whether individuals meet a minimum criteria necessary for inclusion in an FAI population. The IdFAI is intended to give both researchers and clinicians a simple and effective tool to determine an individual's ankle stability status

SUMMARY:
Testing the validity and reliability of IdFAI

DETAILED DESCRIPTION:
reliability & validity of Identification Functional Ankle Instability Questionnaire (IdFAI) Arabic version were assessed in reference to Lower Extremity Functional Scale among repeated ankle sprains college students in Cairo. These college students were randomly selected from different colleges in Cairo University

ELIGIBILITY:
Inclusion Criteria:

* eighty six male and female college students will voluntarily participate in the study

Exclusion Criteria:

* Previous ankle surgery.
* History of any ankle surgery.
* History of fracture within the last 6 months.
* Been involved in any previous strengthening or athletic training program.

Ages: 18 Years to 24 Years | Sex: All
Age Groups: Adult
Study Population: male and female college students
Sampling Method: Non-Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2018-03-10 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-01-22 (Actual)

PRIMARY OUTCOMES:
Validity | 3 months
  Correlation coefficient
Reliability | 3 months
  Cronbach's Alpha

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Giza, Egypt